CLINICAL TRIAL: NCT01778946
Title: Nicotinic Treatment of Age-Related Cognitive Decline in Down Syndrome: An Open Label Pilot Trial
Brief Title: Nicotine Treatment of Cognitive Decline in Down Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Paul Newhouse, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121759
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Down Syndrome; Mild Cognitive Impairment
Keywords: Nicotine; Down Syndrome; Mild Cognitive Impairment; Event Related Potential; Memory; Attention; Trisomy 21; Neuroprotection; Cognitive Enhancement; Alzheimer's Disease; Dementia; APOE
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Nicotine; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine (Experimental): Low Dose Nicotine (7mg) Moderate Dose Nicotine (14mg)
  All participants in study will begin with the 7mg patch, titrating from 2 hours/day to a full 16 hours/day over the course of the first 7 days (based on individual tolerance).
  Day 7 - Day 28 of the study, participants will apply a new nicotine patch daily. Depending on tolerance, some participants may increase to the moderate dose (14mg) patch.
  All participants will apply a new patch daily for a total of 28 days (1 month)
  Interventions: Drug: Low Dose Nicotine (7mg); Drug: Moderate Dose Nicotine (14mg)

INTERVENTIONS:
Drug: Low Dose Nicotine (7mg)
  Other Names: Transdermal Nicotine Patch; Nicotine Skin Patch; Adhesive Nicotine Patch
Drug: Moderate Dose Nicotine (14mg)
  Other Names: Transdermal Nicotine Patch; Nicotine Skin Patch; Adhesive Nicotine Patch

SUMMARY:
This study will ascertain whether nicotine is safe and tolerable in DS patients, help with dose-ranging of nicotine in DS, look for evidence of enhancements in cognitive functioning, and establish evidence for biological and behavioral correlates of nicotinic stimulation effects. The knowledge gained from the translational aspects of this project may also guide the application of new nicotinic drugs in DS and generate, for the first time, data on the importance of nicotinic receptor changes in the development of cognitive impairment in DS adults.

Hypotheses:

* Transdermal nicotine treatment will be well tolerated out to one month by non-smoking DS patients without significant adverse effects.
* Nicotine will enhance cognitive performance by one month compared to baseline and post-treatment testing.
* Nicotine will enhance functioning detectable by clinician and/or informant ratings (pre-post).

DETAILED DESCRIPTION:
Over 50% of adults with Down Syndrome (DS) develop Alzheimer's disease (AD) by the age of 60 (Nadel 2003), and life expectancy in DS is now 50-60 years. Thus, age-associated cognitive impairment and dementia in older adults with DS is an urgent public health concern. The investigators propose that nicotinic stimulation is a promising strategy to stabilize or improve cognitive functioning in adults with DS, possibly with additional neuroprotective effects. The investigators have extensive experience investigating the role of nicotinic receptors on human cognition and impairment. This application takes advantage of new insights into treating Mild Cognitive Impairment (MCI-the precursor condition to Alzheimer's Disease (AD) in typically developing individuals) with nicotine to propose an open label pilot study of transdermal nicotine in middle-aged non-smoking DS patients who show early cognitive and/or behavioral changes consistent with MCI/dementia.

The goal of this study is to establish preliminary evidence for safety, gain preliminary evidence as to whether nicotine enhances cognitive functioning in DS adults, and examine electrophysiological, biological, and behavioral correlates of nicotinic stimulation effects.

The investigators propose that positive results on cognitive or functional indices that would lead to a larger and longer double-blind trial to test more definitively whether nicotinic stimulation may be cognitively and/or functionally enhancing for DS patients. The knowledge gained from the translational aspects of this project will guide the development of potentially new nicotinic drugs in DS and generate, for the first time, data on the importance of nicotinic receptor changes in the development of cognitive impairment in DS adults. This work also represents the first time that cutting-edge advances in treating MCI/AD in the general population are immediately and rigorously applied to those with DS.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive complaints and/or memory difficulties which are verified as new onset by an informant.
* Cognitive Global Rating consistent with mild impairment or deterioration from premorbid baseline.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease/dementia cannot be made by the physician at the time of the screening visit.
* No significant cerebrovascular disease: Modified Hachinski score of less than or equal to 4.
* Age 25+.
* Stable medications for at least 1 month prior to screening. Central nervous system (CNS) medications should be stable for 3 months.
* No evidence of major depression.
* Informant is available who has frequent contact with the subject (e.g. an average of 10 hours per week or more).
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Good general health with no additional diseases expected to interfere with the study.
* Normal B12, rapid plasma reagin (RPR), and Thyroid Function Tests or without any clinically significant abnormalities that would be expected to interfere with the study.
* ECG without clinically significant abnormalities that would be expected to interfere with the study.
* Subject is not pregnant, lactating.
* Subjects will be taking no drugs with cholinergic properties (e.g donepezil).
* Agreement not to take other vitamin or supplements other than multivitamins.
* Negative urine pregnancy test in females.

Exclusion Criteria:

* Any significant neurologic disease such as Alzheimer's disease, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* Active Major depression or another major psychiatric disorder as described in DSM-IV.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including:
* History of myocardial infarction in the past year or unstable or severe cardiovascular disease including angina or congestive heart failure (CHF) with symptoms at rest.
* Clinically significant obstructive pulmonary disease or asthma.
* Clinically significant and unstable gastrointestinal disorder such as ulcer disease or a history of active or occult gastrointestinal bleeding within two years.
* Clinically significant laboratory test abnormalities on the battery of screening tests (hematology, chemistry, urinalysis, ECG).
* Insulin-requiring diabetes or uncontrolled diabetes mellitus.
* Uncontrolled hypertension (systolic BP> 170 or diastolic BP> 100).
* Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, MD, Principal Investigator — Vanderbilt University Dept. of Psychiatry; Alexander C Conley, PhD, Study Director — Vanderbilt University Medical Center Dept. of Psychiatry
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for the Vanderbilt Center for Cognitive Medicine — https://www.vumc.org/ccm/
- See also: Website for the Vanderbilt Kennedy Center for research concerning developmental disabilities — https://vkc.vumc.org/vkc/
- See also: Website for the Down Syndrome Association of Middle Tennessee — http://www.somethingextra.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine: Low Dose Nicotine (7mg) Moderate Dose Nicotine (14mg)
  All participants in study will begin with the 7mg patch, titrating from 2 hours/day to a full 16 hours/day over the course of the first 7 days (based on individual tolerance).
  Day 7 - Day 28 of the study, participants will apply a new nicotine patch daily. Depending on tolerance, some participants may increase to the moderate dose (14mg) patch.
  All participants will apply a new patch daily for a total of 28 days (1 month)
  Low Dose Nicotine (7mg)
  Moderate Dose Nicotine (14mg)
Period: Overall Study
Arm/Group | Nicotine
Started | 7
Completed | 4
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nicotine
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 24.9 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Nicotine Intervention
Description: Maximum transdermal nicotine dosage able to be maintained stably by participants.
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Groups:
- Nicotine: Low Dose Nicotine (7mg) Moderate Dose Nicotine (14mg)
  All participants in study will begin with the 7mg patch, titrating from 2 hours/day to a full 16 hours/day over the course of the first 7 days (based on individual tolerance).
  Day 7 - Day 28 of the study, participants will apply a new nicotine patch daily. Depending on tolerance, some participants may increase to the moderate dose (14mg) patch.
  All participants will apply a new patch daily for a total of 28 days (1 month)
  Low Dose Nicotine (7mg); Moderate Dose Nicotine (14mg)
Arm/Group | Nicotine
Number analyzed (Participants) | 4
Participants
  7 mg | 1
  14 mg | 3

2. Secondary Outcome: Cognitive Improvement - Simple Response Time
Description: Psychomotor speed was measured by the performance on the CANTAB simple reaction time task
Time Frame: 4 time-points over the 6-week testing period: at baseline, day 14, day 28 (end of treatment), and 2-weeks post-treatment on day 42.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Nicotine
Number analyzed (Participants) | 4
ms
  Baseline | 760.08 (542.96)
  Day 14 | 737.13 (566.94)
  Day 28 | 695.52 (344.87)
  Day 42 | 772.79 (552.51)

3. Secondary Outcome: Exploratory - Event-Related Potentials
Description: The investigators will measure daily low-moderate dose nicotine treatment's changes to electrophysiological markers of memory performance using an incidental memory task. The incidental memory task consists of presenting participants with a series of 60 complex images, 50 of which are presented once, and 10 which are repeated 5 times each. The task measures the presence of the late positive potential (LPP), a positive deflection over the parietal cortex which is elevated for the repeated compared to the singly presented images. The presence of this potential is indicative of improved recognition memory.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Nicotine
Number analyzed (Participants) | 4
µV
  Baseline Repeated | 7.95 (0.78)
  Day 14 Repeated | 6.64 (5.44)
  Day 28 Repeated | 6.64 (4.8)
  Day 42 Repeated | 7.49 (3.1)
  Baseline Single | 6.87 (2.03)
  Day 14 Single | 6.76 (2.38)
  Day 28 Single | 5.83 (3.3)
  Day 42 Single | 5.09 (1.33)

4. Secondary Outcome: Cognitive Improvement - Continuous Performance Test
Description: Performance on the Conners' Continuous Performance Test, which is a measure of sustained attention. The main outcome measure was commission errors, which measures attention failures. The commission errors are calculated as T-scores. Higher T-scores indicate worse performance, lower T-scores indicate better performance. Average performance is a score of 50, with a standard deviation of 10.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Nicotine
Number analyzed (Participants) | 4
T-score
  Baseline | 47.82 (11.46)
  Day 14 | 49.23 (6.41)
  Day 28 | 43 (7.41)
  Day 42 | 42.95 (8.2)

5. Secondary Outcome: Cognitive Improvement - Buschke Selective Reminding Task
Description: Episodic memory performance was assessed by the Buschke Selective Reminding Task. The main outcome metric of this test was the total words correctly recalled.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Words Correctly Recalled
Arm/Group | Nicotine
Number analyzed (Participants) | 4
Words Correctly Recalled
  Baseline | 33.75 (24.42)
  Day 14 | 41.5 (30.97)
  Day 28 | 54.5 (33.89)
  Day 42 | 45.5 (32.72)

6. Secondary Outcome: Cognitive Improvement - Critical Flicker Fusion Task
Description: Arousal and vigilance were measured by the Critical Flicker Fusion task. The task used at perceptual performance on ascending and descending frequencies of the task.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Nicotine
Number analyzed (Participants) | 4
Hz
  Baseline Ascending Frequency | 20.6 (8.7)
  Day 14 Ascending Frequency | 29.7 (8.4)
  Day 28 Ascending Frequency | 31.6 (8.27)
  Day 42 Ascending Frequency | 30 (11.7)
  Baseline Descending Frequency | 36.9 (9.01)
  Day 14 Descending Frequency | 31.3 (4.23)
  Day 28 Descending Frequency | 26.3 (6.51)
  Day 42 Descending Frequency | 26.2 (4.65)

ADVERSE EVENTS:
Time Frame: 6-weeks
Description: Adverse events collected through query of subjects about any new or worsening problems or side effects, conducted at each contact.
Arm/Group | Nicotine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine (N=7)
Nausea (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT01778946/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT01778946/ICF_001.pdf